CLINICAL TRIAL: NCT02035098
Title: The Effectiveness of the Quality Program Pac-IficO to Improve Pain Management in Hospitalized Cancer Patients. A Before-after Cluster Phase II Trial
Brief Title: Improving Pain Management in Hospitalized Cancer Patients. A Before-after Cluster Phase II Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RFPS-2006-6-341684
Record Dates: First submitted 2013-11-08; First posted 2014-01-14 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2013-11

CONDITIONS: Cancer
Keywords: cancer, pain, cluster trial, quality improvement
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The Pac-IFicO programme (Experimental): The Pac-IFicO programme is a complex interventions aimed at improving the quality of pain managementi in hospitalized patients.
  Interventions: Other: the Pac-IFicO programme

INTERVENTIONS:
Other: the Pac-IFicO programme — The Pac-IFicO programme is a complex interventions with multiple components. It includes focus group with ward professionals for identifying possible local obstacles to optimal pain control, informative material for the patients, an educational programs performed through guides from the wards, and an organisational intervention to the ward.

SUMMARY:
The objective of the study is to evaluate the efficacy of the Pac-IFicO programme in improving the quality of pain management in hospitalised cancer patients. This is a before-after cluster phase II study performed in medicine, oncology and respiratory disease hospital wards. The Pac-IFicO programme is a complex interventions with multiple components. The primary end-point of the study is the proportion of cancer patients with severe pain.

DETAILED DESCRIPTION:
Cancer-related pain continues to be a major healthcare issue worldwide. Despite the availability of effective analgesic drugs, published guidelines and educational programs for Health Care Professionals the symptom is still under-diagnosed and its treatment is not appropriate in many patients.

The objective of the study is to evaluate the efficacy of the Pac-IFicO programme in improving the quality of pain management in hospitalised cancer patients.

This is a before-after cluster phase II study. After the before assessment, the Pac-IFicO programme will be implemented in ten medicine, oncology and respiratory disease hospital wards. The same assessment will be repeated after the completion of the intervention.

The Pac-IFicO programme is a complex interventions with multiple components. It includes focus group with ward professionals for identifying possible local obstacles to optimal pain control, informative material for the patients, an educational programs performed through guides from the wards, and an organisational intervention to the ward.

The primary end-point of the study is the proportion of cancer patients with severe pain. Secondary end-points include opioids administered in the wards, knowledge in pain management, quality of pain management. We plan to recruit about 500 cancer patients from ten hospital wards. This sample size should be sufficient, after appropriate statistical adjustments for clustering, to detect an absolute decrease in the proportion of cancer patients with severe pain (the primary end-point) from 20% to 9%.

ELIGIBILITY:
Inclusion criteria

WARD LEVEL

1. consent from the head of the ward to participate to the study;
2. ward classified as oncology, medicine, respiratory disease ward according to the regional classification of hospitals;
3. number of beds: ≥20 ;
4. number of ordinary admissions with primary or secondary diagnosis of tumour (ICD-IX 140-239) >180 per year;
5. yearly average stay in hospital between 4 and 19 days;
6. punctual prevalence of patients with primary or secondary diagnosis of tumour (ICD-IX 140-239) ≥ 8 patients.

STAFF LEVEL

1. affiliation to the ward;
2. informed consent to participate to the study.

PATIENT LEVEL

1. ordinarily admitted in the ward for at least 24 hours;
2. age ≥ 18 years
3. able to fill in the questionnaire according the profession judgment;
4. informed consent to participate to the study.

Exclusion criteria

WARD LEVEL

1. the ward had received or is receiving quality improvement programme of staff education for improve pain control.

PATIENT LEVEL

1. patient already assessed in one of the previous assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
percentage of hospitalized cancer patients with average severe pain (score 7-10) within the latest 24 hours | up to 28±1 days after Pac-IficO completion.
  All eligible patients will be assessed in the month before (the before sample) and in the month after the implementation of the intervention (the after sample). For both samples the outcomes are composite measures from the five assessments in the month before and from five assessments in the month after. Each outcome results from the sum of patients with severe pain in the five assessments (the numerator) divided the total number of assessed patients in the five assessments (the denominator) x 100.

SECONDARY OUTCOMES:
knowledge of the ward professionals in pain management | In the month before and in the month after the completion of the intervention.
  Knowledge of the ward professionals in pain management were assessed before and after the implementation of the intervention by administering the Italian version of the Pain Attitudes and Knowledge Scale (PAK)
quality of pain management in cancer patients | up to 28±1 days after Pac-IficO completion
  All eligible patients will be assessed in the month before (the before sample) and in the month after the implementation of the intervention (the after sample). For both samples the outcomes are composite measures from the five assessments in the month before and from five assessments in the month after. Each outcome results from the sum of patients with severe pain in the five assessments (the numerator) divided the total number of assessed patients in the five assessments (the denominator) x 100.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Peruselli, MD, Principal Investigator — ASL Biella (Italy)

REFERENCES:
- [Derived] Ripamonti CI, Prandi C, Costantini M, Perfetti E, Pellegrini F, Visentin M, Garrino L, De Luca A, Pessi MA, Peruselli C. The effectiveness of the quality program Pac-IficO to improve pain management in hospitalized cancer patients: a before-after cluster phase II trial. BMC Palliat Care. 2014 Mar 29;13(1):15. doi: 10.1186/1472-684X-13-15. PMID 24678911